CLINICAL TRIAL: NCT05255211
Title: Effect on Early Cognition Under Sedation by Rimazole Toluenesulfonate in Old Patient Undergoing Colonoscopy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WanYi（2020-5）
Record Dates: First submitted 2021-12-02; First posted 2022-02-24 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Cognition
Keywords: Remimazolam tosilate; cognition; Old; Colonoscopy
MeSH Terms: interventions — Propofol; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Remimazolam (Experimental): IV Remimazolam tosilate 0.3mg/kg
  Interventions: Drug: Remimazolam tosilate
- propofol (Active Comparator): IV propofol 1.2~2.5mg/kg
  Interventions: Drug: Propofol
- saline (Placebo Comparator): IV saline solution 10ml
  Interventions: Other: saline solution

INTERVENTIONS:
Drug: Remimazolam tosilate — IV before procedure
  Other Names: experimental
  Arms: Remimazolam
Drug: Propofol — IV before procedure
  Other Names: active comparator
  Arms: propofol
Other: saline solution — IV before procedure
  Other Names: placebo comparator
  Arms: saline

SUMMARY:
To investigate the effect on cognition under sedation by Rimazole toluenesulfonatein elderly patients undergoing colonoscopy

ELIGIBILITY:
Inclusion Criteria:

1. ASA I~II
2. patients will be treatmented by sedation under colonoscopy
3. sign informed consent

Exclusion Criteria:

(1) Preoperative depression and cognitive impairment

（2） Hearing or visual impairment;

（3） Drug abuse, alcoholism or long-term use of antidepressants;

（4） Cardiovascular and cerebrovascular accidents, neurological sequelae, or severe liver and kidney function damage occurred within 6 months

（5） BMI < 18, BMI > 30

（6） Confirmed or suspected allergy to the test drug

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-12-02 (Actual); Primary Completion 2024-12-02 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Mini-mental State Examination(MMSE) score 1 | 5 minutes before procedure
  The MMSE scoring standard is the preferred scale for dementia screening. It can comprehensively, accurately and quickly reflect the mental state and cognitive defects of the subjects.The values is 0~30.
  Cognitive dysfunction: the highest score is 30 points, the score is normal at 27-30, and the score <27 is cognitive dysfunction; Dementia classification criteria: illiteracy ≤ 17, primary school level ≤ 20, secondary school level (including technical secondary school) ≤ 22 points, university level (including junior college) ≤ 23 points; 3. Dementia severity classification: mild MMSE ≥21 points; moderate, MMSE 10-20 points; severe, MMSE ≤9 points;
Mini-mental State Examination(MMSE) score 2 | 30 minutes after colonoscopy when VAAS score>=4
  The MMSE scoring standard is the preferred scale for dementia screening. It can comprehensively, accurately and quickly reflect the mental state and cognitive defects of the subjects.The values is 0~30.
  Cognitive dysfunction: the highest score is 30 points, the score is normal at 27-30, and the score <27 is cognitive dysfunction; Dementia classification criteria: illiteracy ≤ 17, primary school level ≤ 20, secondary school level (including technical secondary school) ≤ 22 points, university level (including junior college) ≤ 23 points; 3. Dementia severity classification: mild MMSE ≥21 points; moderate, MMSE 10-20 points; severe, MMSE ≤9 points;

CONTACTS AND LOCATIONS:
Locations (1):
- Yongming Chen, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No